CLINICAL TRIAL: NCT01895660
Title: A Multisite Trial of Pediatric Constraint-Induced Movement Therapy
Brief Title: Children With Hemiparesis Arm and Hand Movement Project (CHAMP Study)
Acronym: CHAMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Ohio State University (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Stephanie DeLuca, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1RO11HD068345-01A1
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Hemiparesis; Cerebral Palsy; Brain Injury
Keywords: P-CIMT; Pediatric Constraint Induced Movement Therapy; Hemiparesis; Cerebral Palsy; Children
MeSH Terms: conditions — Paresis; Cerebral Palsy; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group with continuous constraint and daily therapy (Experimental)
  Interventions: Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation
- Group with continuous constrainit and 3 days a week therapy (Experimental)
  Interventions: Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation
- Group with part-time constraint and daily therapy (Experimental)
  Interventions: Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation
- Group with part-time constraint and 3 days a week therapy (Experimental)
  Interventions: Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation
- Usual and customary treatment group (Active Comparator)
  Interventions: Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation

INTERVENTIONS:
Behavioral: Variations in Pediatric Constraint-Induced Movement Therapy (P-CIMT) versus usual and customary rehabilitation — Types of constraint and dosage amounts will be varied.

SUMMARY:
What is the CHAMP Study?

The CHAMP Study is a multisite clinical trial funded by the National Institutes of Health that is comparing the efficacy of alternative therapies for young children with unilateral spastic cerebral palsy (or hemiparetic cerebral palsy). Children who meet study eligibility criteria at one of the three clinical sites (Roanoke, VA; Charlottesville, VA, and Columbus, OH) will be invited to enroll, and their parents will be provided all necessary paperwork along with informed consent documentation. Assignment to one of the alternative therapy conditions will be random. Participation in the study includes assessment of each child prior to treatment, close monitoring of the child's progress during treatment, and post-treatment evaluation at the end of therapy, as well as, 6 and 12 months later. Parents will have an active role in the project, both observing their child during therapy sessions and then engaging in home-based activities that allow the child to practice and extend new motor skills. There will be no charge for the therapy provided.

What are the therapies being tested? In the past decade or so, a new form of therapy for children with hemiparetic cerebral palsy was developed and has shown to produce positive changes in individual children and in small clinical trials (e.g., DeLuca, Echols, Ramey, & Taub, 2003; DeLuca, Echols, Law, & Ramey, 2006; Case-Smith, DeLuca, Stevenson, & Ramey, 2012). The therapy is named Constraint-Induced Movement Therapy (CIMT) and refers to a multi-component form of therapy in which the child has the unimpaired or less impaired upper extremity constrained (by a cast or a splint) while also receiving active therapy from a specially trained therapist who shapes new skills and functional activities with the child's more impaired upper extremity. Traditionally, CIMT therapy dosages have been high - often lasting many hours per day, 5 days a week, for 4 consecutive weeks. There are important clinical and scientific questions that need to be answered about the effects of different dosage levels and about different types of constraint on the child's more functional (less impaired) arm and hand. This study will be the first that will directly compare different amounts of therapy and different types of constraint to evaluate what "works best" for young children. The therapy is very play-like and engaging for children, and no negative effects of casting or the high dosages have been detected in previous clinical trials.

Who is eligible: Children between 2 and 8 years of age with a diagnosis of unilateral spastic cerebral palsy or hemiparetic cerebral palsy. Children must be relatively healthy, not currently receiving Botox (or other similar medications), and able to understand simple communication and instructions. In advance, the treatment will be explained in detail to parents and a written protocol available to share with the child's physician and other current therapist for review. During the one month of treatment, children will not receive other forms of physical or occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

1. are 2 years - 8 years old
2. do not have any serious complicating conditions or acute medical concerns
3. are diagnosed with cerebral palsy with hemiparesis (prior to age 2)
4. have not had botox injections in the last 6 months and
5. have not received Constraint-Induced Movement Therapy in the last 6 months
6. have a clinical MRI that can be provided in digital format for research project

Exclusion Criteria:

-

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2013-07; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Functional measurements of change across time in the child's abilities with their arms and hands will be measured using the Assisting Hand Assessment, the Peabody Developmental Motor Scales, and the Pediatric Evaluation and Disability Inventory. | Pretreatment; Post-Treatment, 6 and 12 months Follow up
  Functional measurements of arm use

SECONDARY OUTCOMES:
Modified version of Quality of Upper Extremity Skills Test (QUEST) | Pre treatment; Post-Treatment (end of 4 weeks of treatment), 6 and 12 months Follow up
  Functional range of motion measure

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech, Roanoke, Virginia, United States

REFERENCES:
- [Derived] Ramey SL, DeLuca SC, Stevenson RD, Conaway M, Darragh AR, Lo W; CHAMP. Constraint-Induced Movement Therapy for Cerebral Palsy: A Randomized Trial. Pediatrics. 2021 Nov;148(5):e2020033878. doi: 10.1542/peds.2020-033878. Epub 2021 Oct 14. PMID 34649982
- [Derived] Ramey SL, DeLuca S, Stevenson RD, Case-Smith J, Darragh A, Conaway M. Children with Hemiparesis Arm and Movement Project (CHAMP): protocol for a multisite comparative efficacy trial of paediatric constraint-induced movement therapy (CIMT) testing effects of dosage and type of constraint for children with hemiparetic cerebral palsy. BMJ Open. 2019 Jan 15;9(1):e023285. doi: 10.1136/bmjopen-2018-023285. PMID 30782701